CLINICAL TRIAL: NCT05766631
Title: Treating Polysubstance Use in Methadone Maintenance: Application of Novel Digital Technology
Brief Title: Treating Polysubstance Use Using a Novel Digital Technology
Acronym: POLY
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Friends Research Institute, Inc. (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 11387; 1R01DA057608-01 (NIH)
Record Dates: First submitted 2023-02-24; First posted 2023-03-13 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Opioid Use; Opioid Use Disorder; Cocaine Use; Cocaine Use Disorder
Keywords: methadone; telehealth; mHealth; medications for opioid use disorder (MOUD)
MeSH Terms: conditions — Opioid-Related Disorders

STUDY DESIGN:
Intervention Model Description: Two-arm, parallel random assignment (covariate-adaptive allocation to ensure equal distribution of three variables across groups: age, gender, recent cocaine use) with assessments at baseline, as well as 3-/6-/12-months post randomization.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Methadone Treatment-as-Usual (Active Comparator): Participants randomized to the Methadone Treatment-as-Usual (TAU) Condition will receive treatment-as-usual at the community methadone clinics, which will include daily medication, individual and group addiction counseling, and outpatient or intensive outpatient behavioral health services, depending on the clinic and the needs of the patient. After randomization into the TAU arm, participants will complete the program's psychosocial and medical intake, methadone dose induction and adjustment, and provide urine tests and receive medication take-homes per the program's policies and methadone treatment regulations.
  Interventions: Drug: Methadone Treatment-As-Usual
- DynamiCare Plus Methadone Treatment-as-Usual (Experimental): DynamiCare Plus Methadone Treatment-as-Usual (DCM+TAU) participants will receive the same services as TAU participants, plus access to the DynamiCare Health smartphone app for 48 weeks. After randomization, the research assistant (RA) will download the DynamiCare Health app onto their smart phone (or provide them with a smartphone with the app already installed). Participants will get oral fluid testing kits and a Next Step debit card. Participants will be trained in use of the app and oral fluid test kits and will practice until they can produce two valid tests in a row without aid of the research staff. Participants will earn $40 for successful completion of the orientation and training. DCM+TAU participants will then use the app to complete remote random drug screenings, prove attendance to appointments and medication pickups, interact with modules designed to improve substance use reductions, and other treatment-related activities.
  Interventions: Behavioral: DynamiCare Health; Drug: Methadone Treatment-As-Usual

INTERVENTIONS:
Behavioral: DynamiCare Health — Participants earn incentives for:
  1. CM for opioid and cocaine abstinence. Accomplished via oral fluid (saliva) test kits given to participants.
  2. Patients who test negative on opioids and cocaine are also eligible for a bonus if they additionally test negative for non-targeted drugs (except methadone).
  3. Patients will receive notices of their medication pickup appointments through the app itself, and monetary rewards will be delivered to the Next Step debit card when the participant's presence at the clinic is verified by clinic records.
  4. The app provides 72 self-administered modules based on the principles of cognitive behavioral therapy that are designed to aid in relapse prevention; small incentive rewards ($1) are provided for completion of up to 3 modules per week for the first weeks of treatment.
  Other Names: DCH
  Arms: DynamiCare Plus Methadone Treatment-as-Usual
Drug: Methadone Treatment-As-Usual — Participants will receive treatment-as-usual at the methadone clinic, including daily methadone dosing, individual and group addiction counseling, and OP or IOP behavioral health services, depending on the clinic and the needs of the patient.

SUMMARY:
The goal of this clinical trial is to determine the effects of an app to reduce opioid and cocaine use when layered atop methadone treatment as usual among people using both opioids and cocaine. The main questions it aims to answer are:

* Do people who use the app remain in methadone treatment longer than people who receive only treatment as usual?
* Do people who use the app report using opioids and/or cocaine less often, and do they report better improvements in their quality of life, than people who receive only treatment as usual?
* Does using the app more lead to better methadone treatment outcomes among people using the app?

Participants in this study will be randomly assigned to receive either the app or methadone treatment as usual. Participants randomly assigned to the treatment as usual group will receive access to methadone services as normally provided, including scheduled access to medications, information about the consequences of opioid and other drug use, and any onsite services (including group based interventions and/or 12-step programs). Those randomized into the app-using group will receive all the same services as the treatment as usual group, but will also be given a phone with the app already installed, or will have the app installed on their existing phone if they already have one. At random times throughout the week, the app will ask participants to submit drug tests for opioids and cocaine, which participants will be able to do remotely without having to physically "go to" a testing site. For each test that demonstrates the participant hasn't used opioids or cocaine, the participant will be rewarded with money directly into a debit card. Participants will also be able to earn rewards for picking up treatment-related medications, attending onsite appointments, and other treatment-related activities.

DETAILED DESCRIPTION:
This two-arm randomized trial will evaluate the impact of 48 weeks of the DynamiCare app-based CM (DCM) intervention on retention in methadone treatment and polysubstance use among 240 methadone maintenance (OTP) patients with comorbid opioid use disorder and cocaine use disorder. New enrollees in methadone maintenance at two community treatment programs will be randomly assigned to either methadone treatment-as-usual (TAU) at the OTP or methadone TAU paired with the DynamiCare Health app (TAU+DCM) including remote drug testing and monetary rewards for negative opioid and cocaine tests indicating abstinence. Data on methadone treatment retention will be obtained through OTP records, and follow-up assessments will be conducted at 3-, 6-, and 12-months post-enrollment.

The study will examine participant outcomes in the domains of three aims:

Aim 1: To determine the relative effectiveness of TAU+DCM compared to TAU alone in improving methadone treatment retention through 12-months post treatment entry.

Aim 2: To determine the relative effectiveness of TAU+DCM compared to TAU alone in terms of [AIM 2a] reducing opioid use and cocaine use; and [Aim 2b] improving other secondary outcomes including non-targeted substance use and quality of life through 12-months post treatment entry.

Aim 3: To explore app use patterns, acceptability, and perceived value of personalized content on opioid and polysubstance use through 12-months post treatment entry.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 or older
2. Cocaine use (self-reported in the past 30 days)
3. Willing and able to provide informed consent

Exclusion Criteria:

1. Severe psychiatric disorders
2. On home detention
3. Visual impairment that would make the use of the phone app impractical
4. Living arrangement that currently restricts phone access

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2023-07-26 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-09-29 (Estimated)

PRIMARY OUTCOMES:
Retention in Methadone Treatment through 48 Weeks | 48 weeks
  The primary outcome of the proposed study is retention in methadone treatment, which will be determined via clinic attendance records, and will be defined as 7 days of continuous absence from scheduled clinic medication visits at any point during the 48-week intervention period.

SECONDARY OUTCOMES:
Drug Use through 48 Weeks | 48 weeks
  Self-reported data, clinical records, urinalysis at baseline and 3-/6-/12-month follow-ups, as well as random drug testing associated with the DynamiCare app will all be used in concert to determine opioid, cocaine, and other drug use during the 48-week intervention period.
Changes in Quality of Life through 48 Weeks | 48 weeks
  Self-report data collected at baseline as well as at the 3-/6-/12-month follow-up assessments will assess changes in participants quality of life, including familial, legal, and/or medical issues, during the 48-week intervention period.

CONTACTS AND LOCATIONS:
Overall Officials: Karen Alexander, Ph.D., Principal Investigator — Friends Research Institute, Inc.
Locations (5):
- United States (5):
  - Friends Research Institute, Inc. Central Office, Baltimore, Maryland
  - Glenwood Life Counseling Center, Baltimore, Maryland
  - Institutes for Behavior Resources, Baltimore, Maryland
  - Man Alive, Baltimore, Maryland
  - BD Health Services, Inc. -- Dundalk, Baltimore, Maryland

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Alexander K, Sharma A, Fletcher JB, Smith Z, Huddleston T, Gryczynski J, Stitzer M. Digitally delivered contingency management during methadone treatment for people with co-occurring cocaine and opioid use: a protocol for a randomized controlled trial. Front Psychiatry. 2025 Jul 2;16:1576277. doi: 10.3389/fpsyt.2025.1576277. eCollection 2025. PMID 40673228